CLINICAL TRIAL: NCT02323490
Title: Augmentation of Meniscal Repair With Bone Marrow Stimulation Techniques (Microfractures): a Double Blind, Prospective, Randomized Clinical Trial of Efficacy and Safety.
Brief Title: Augmentation of Meniscal Repair With Marrow Stimulation Techniques (Microfractures)
Acronym: men_micro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Rafał Kamiński, M.D. Ph.D., Centre of Postgraduate Medical Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: men_micro
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Meniscus Lesion
Keywords: meniscus repair; bone marrow stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- with microfractures (Experimental): Standardized meniscal repair with bone marrow stimulation techniques (microfractures)
  Interventions: Procedure: with microfractures
- without microfractures (Placebo Comparator): Standardized meniscal repair without augmentation
  Interventions: Procedure: without microfractures

INTERVENTIONS:
Procedure: with microfractures — following meniscal repair, microfractures will be created on the intercondylar and outer part of femoral condyle (outside of joint surface), lateral or medial, respectively
  Arms: with microfractures
Procedure: without microfractures — standard procedure meniscal repair without augmentation.
  Arms: without microfractures

SUMMARY:
This study will compare meniscal healing augmented or without augmentation with bone marrow stimulation techniques The assessments will include validated, disease specific, patient oriented outcome measures, second look arthroscopy during second step ACL reconstruction. Results of this study will help ascertain whether microfractures improve meniscal healing rates.

DETAILED DESCRIPTION:
The role of meniscal in the knee integrity is pivotal and lack or partial role of the meniscus increases rate of joint degeneration. Partial meniscal removal is the most popular procedure and meniscal repair remain in minority of arthroscopic surgeries. As criteria of inclusion to meniscal repair are very rough, still success rates of meniscal repair remain in the 60-80% range for isolated repairs. This rate is greater when performed with ACL reconstruction. We believe that augmentation with bone marrow stimulation techniques will induce more complete and possibly faster healing.

ELIGIBILITY:
Inclusion Criteria:

* Complete vertical longitudinal tear > 10 mm in length
* Tear located in the vascular portion of the meniscus, only in red-white zone
* Unstable peripheral tear
* Single tear of the medial and/or lateral meniscus
* Meniscal injury 1 -18 month prior surgery
* Planned second step arthroscopy (ACL reconstruction)
* Skeletally mature patients 18-55 years of age

Exclusion Criteria:

* discoid meniscus
* arthritic changes (Kellgren Lawrence scale >2)
* non repairable meniscus
* degenerative or presence of crystals in meniscus
* concomitant procedure (acl reconstruction, microfracturing, trephination)
* inflammatory diseases (i.e. rheumatoid arthritis)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08-19 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Second look arthroscopy (assessment of meniscal healing integrity during second look) | 8-18 weeks
  The primary outcome measures will be assessment of meniscal healing integrity during second look arthroscopy 3-5 months post repair.

SECONDARY OUTCOMES:
Visual Analog Scale | 6 weeks, 12 weeks, 6mts, 1yr post op, 2yrs post op, 3 yrs post op
  Pain Visual Analog Scale.
Knee injury and Osteoarthritis Outcome Score scale | 6 weeks, 12 weeks, 6mts, 1yr post op, 2yrs post op, 3 yrs post op
  Knee injury and Osteoarthritis Outcome Score
International Knee Documentation Committee - Subjective Knee Evaluation Form | 6 weeks, 12 weeks, 6mts, 1yr post op, 2yrs post op, 3 yrs post op
  International Knee Documentation Committee - Subjective Knee Evaluation Form
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 weeks, 12 weeks, 6mts, 1yr post op, 2yrs post op, 3 yrs post op
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Kamiński, M.D. Ph.D., Principal Investigator — SPSK Prof A. Gruca Hospital
Locations (1):
- Prof. A. Gruca Teaching Hospital, The Medical Centre of Postgraduate Education, Otwock, Woj. Mazowieckie, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kaminski R, Kulinski K, Kozar-Kaminska K, Wasko MK, Langner M, Pomianowski S. Repair Augmentation of Unstable, Complete Vertical Meniscal Tears With Bone Marrow Venting Procedure: A Prospective, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study. Arthroscopy. 2019 May;35(5):1500-1508.e1. doi: 10.1016/j.arthro.2018.11.056. Epub 2019 Mar 20. PMID 30902532